CLINICAL TRIAL: NCT04425447
Title: Thoracic Interfascial Plane Block Versus Thoracic Paravertebral Block for Anesthesia in Gynecomastia Surgery: A Randomized Controlled Trial
Brief Title: Thoracic Interfascial Plane Block Versus Thoracic Paravertebral Block in Gynecomastia Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Taysser Mahmoud Abdalraheem, Principal Investigator - Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 33793/4/20
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Gynecomastia; Thoracic Interfascial Plane Block; Thoracic Paravertebral Block; Anesthesia
MeSH Terms: conditions — Gynecomastia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Active Comparator): 30 patients will receive bilateral tumescent local anesthesia as a control group
  Interventions: Drug: Tumescent local anesthesia
- Group TPVB (Experimental): 30 patients will receive bilateral US guided thoracic paravertebral block.
  Interventions: Drug: Thoracic paravertebral block
- Group TIPB (Experimental): 30 patients will receive bilateral US guided thoracic interfascial plane block
  Interventions: Drug: Thoracic interfascial plane block

INTERVENTIONS:
Drug: Tumescent local anesthesia — Surgical disinfection of the area will be performed, skin inﬁltration with 2 mL of 1% lidocaine will be done, and wetting fluid will be used (1000 ml normal saline, 20 ml lidocaine 2%, and 1 mg epinephrine).
  Infiltration will be initiated with a 25-gauge needle. The 25-gauge needles cause little discomfort and provide enough local anesthesia to allow painless, more complete infiltration using a 20-gauge spinal needle. After the glandular nipple tissue is made somewhat tumescent, a larger (20-gauge) spinal needle can be more easily passed through the otherwise dense and resistant tissue.
  Arms: Group C
Drug: Thoracic paravertebral block — The paravertebral block (PVB) will be performed in the sitting position. Surgical disinfection of the thoracic paravertebral area will be done. A linear high-frequency transducer will be used. The scanning process (longitudinal out-of-plane technique) will be started at 5 to 10 cm lateral to the spinous process to identify the rounded ribs and parietal pleura underneath. The transducer is then moved progressively more medially until transverse processes are identiﬁed as more squared structure and deeper to the ribs. Once the transverse processes will be identiﬁed, skin inﬁltration with 2 mL of 1% lidocaine will be done. A 100-mm, 22 G needle will be inserted out of the plane to contact the transverse process and then walk off the transverse process 1 to 1.5 cm deeper searching for loss of resistance to inject 20 mL (5mL lidocaine 2% and 15 mL bupivacaine 0.25%) at each level of T4.
  Arms: Group TPVB
Drug: Thoracic interfascial plane block — Total LA injected was 80 mL (10 mL lidocaine 2% and 70 mL bupivacaine 0.25%) The linear probe will be placed below the outer third of the clavicle to detect anatomical landmarks, such as the serratus anterior muscle (SAM), external intercostal muscle (EIM), pectoralis muscles, thoracoacromial artery, and second rib. A test bolus of 1-2 ml of LA will be injected; upon confirmation of diffusion of the test dose between the external intercostal muscles and the SAM, a total of 20 ml of LA will be injected. The needle will be then carefully moved in the direction of the third and fourth ribs while confirming the expansion of the fascial plane.
  In the performance of the pecto-intercostal fascial plane block (PIFB), a probe will be placed parallel to the long axis of the sternum at a distance greater than 2 cm from the attachment of the second rib and sternum to identify the pectoralis muscles, EIM, and second rib. A
  Arms: Group TIPB

SUMMARY:
The growing increase in the number of gynecomastia surgeries has resulted in an increased need for anesthetic techniques with improved pain reduction, safety, and fewer complications.

The aim of this work is to compare the efficacy of ultrasound guided thoracic interfascial plane block and ultrasound guided thoracic paravertebral block for anesthesia in gynecomastia surgery.

DETAILED DESCRIPTION:
This prospective randomized open label clinical trial will be carried out on 90 male patients undergoing elective idiopathic gynecomastia surgery in Tanta University Hospitals.

Study design:

Patients will be randomly allocated into three equal groups by computer generated sequence through sealed opaque envelopes:

Group C: 30 patients will receive bilateral tumescent local anesthesia as a control group.

Group TPVB: 30 patients will receive bilateral US guided thoracic paravertebral block.

Group TIPB: 30 patients will receive bilateral US guided thoracic interfascial plane block.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 up to 65 years
* Male gender only
* ASA physical status I and II
* Weight 75-100 kg
* Duration of surgery ≤ 2 hours
* Scheduled for elective idiopathic gynecomastia surgery

Exclusion Criteria:

* Patient refusal.
* Uncooperative patients.
* Known hypersensitivity to local anesthetic (LA) (bupivacaine).
* Local infection at the site of injection (TPVB or TIPB).
* Coagulopathy.
* History of opioid abuse or chronic analgesic use.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynecomastia in males only
Enrollment: 90 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The amount of intraoperative fentanyl requirement (mg) | 3 hours
  If the patient complains from pain, fentanyl 25μg intravenously will be administrated.

SECONDARY OUTCOMES:
Degree of patient's satisfaction | 6 hours
  Patient satisfaction before discharge using a 5- point score, with (0 = very dissatisfied, 1 = dissatisfied, 2 = neither satisfied nor dissatisfied, 3 = satisfied and 4 = very satisfied).

OTHER OUTCOMES:
Amount of postoperative analgesic requirement (mg) | 24 hours
  Postoperative pain will be assessed by numeric rating scale (NRS) score and diclofenac sodium 75 mg intramuscular will be given as rescue analgesia if NRS score was >3 (maximum 75 mg/8 hours).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, ElGharbiaa, Egypt

IPD SHARING:
Plan to Share IPD: No